CLINICAL TRIAL: NCT01745367
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Study Comparing Tivozanib Hydrochloride in Combination With Paclitaxel v Placebo in Combination With Paclitaxel in Locally Recurrent and/or Metastatic Triple Negative Breast Cancer
Brief Title: Tivozanib in Combination With Paclitaxel in Patients With Locally Recurrent or Metastatic Triple Negative Breast Cancer
Acronym: BATON-BC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV-951-12-204; 2012-003507-35 (EudraCT Number)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Triple Negative Breast Cancer
Keywords: Tivozanib hydrochloride; triple negative breast cancer; paclitaxel; pharmacokinetics; biomarkers; metastatic breast cancer; mBC; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — tivozanib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo in combination with paclitaxel (Active Comparator): Placebo orally once daily on a 3 weeks on/1 week off schedule with 90 mg/m2 of paclitaxel administered intravenously 3 weeks on (Day 1, Day 8 and Day 15)/1 week off (4 weeks = 1 Cycle).
  Interventions: Drug: paclitaxel; Drug: Placebo
- Tivo in combination with paclitaxel (Experimental): 1.5 mg tivozanib hydrochloride orally once daily on a 3 weeks on/1 week off schedule with 90 mg/m2 of paclitaxel administered intravenously 3 weeks on (Day 1, Day 8 and Day 15)/1 week off (4 weeks = 1 Cycle).
  Interventions: Drug: Tivozanib Hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: Tivozanib Hydrochloride
  Other Names: Tivozanib
  Arms: Tivo in combination with paclitaxel
Drug: paclitaxel
  Other Names: PTX
Drug: Placebo
  Arms: Placebo in combination with paclitaxel

SUMMARY:
This is a phase 2 multicenter, double-blind, randomized, placebo-controlled, two-arm study for subjects with locally recurrent or metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
This is a phase 2 multicenter, double-blind, randomized, placebo-controlled, two-arm study for subjects with locally recurrent or metastatic triple negative breast cancer.

Patients will be randomized 2:1 to either tivozanib hydrochloride and weekly paclitaxel or placebo and weekly paclitaxel.

Subjects will be stratified based on Eastern Cooperative Oncology Group (ECOG) performance score (0 vs 1) and line of treatment (first vs second).

All subjects will be evaluated for progression free survival and overall survival as well as safety and tolerability. Biomarker and pharmacokinetic (PK) analysis are also included in study. This study will determine whether tivozanib hydrocholoride combined with weekly paclitaxel improves clinical outcomes in patients with triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally recurrent or metastatic TNBC, defined as ER/PR <1%, HER2 0-1+, or 2+ with negative FISH
* Measurable disease per RECIST version 1.1
* ECOG performance status of 0 or 1
* Confirmed available archival tumor tissue.

Exclusion Criteria:

* More than 1 prior systemic chemotherapy for treatment of locally recurrent or metastatic breast cancer (neoadjuvant and adjuvant therapy is allowed provided the subject did not progress within 12 months of taxane based therapy
* Prior treatment with VEGF pathway targeted agent
* Major surgery within 4 weeks or minor surgery or radiotherapy within 2 weeks of first dose of study drug
* Known history of central nervous system metastasis (subjects with previously treated (radiotherapy or surgery) brain metastasis that have been stable off steroids or enzyme-inducing antiepileptic drugs for at least 3 months following prior treatment may be enrolled)
* Significant hematologic, gastrointestinal, thromboembolic, vascular, bleeding, or coagulation disorders
* Significant serum chemistry or urinalysis abnormalities
* Significant cardiovascular disease, including: uncontrolled hypertension; myocardial infarction or unstable angina within 6 months prior to administration of first dose of study drug; and symptomatic left ventricular dysfunction or baseline left ventricular ejection fraction (LVEF) by multigated acquisition scan (MUGA) or ECHO.
* Severe peripheral neuropathy ≥ Grade 2
* Currently active second primary malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Needle, Study Chair — AVEO Pharmaceuticals, Inc.
Locations (54):
- United States (20):
  - Birmingham, Alabama
  - Jacksonville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Oak Lawn, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Fargo, North Dakota
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Dallas, Texas
  - Galveston, Texas
- Australia (6):
  - Port Macquarie, New South Wales
  - Woodville South, South Australia
  - Bentleigh, Victoria
  - Newcastle
  - South Brisbane
  - St Leonards
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Saint John
- Germany (6):
  - Berlin
  - Cologne
  - Hanau
  - Leipzig
  - Münster
  - Tübingen
- Italy (5):
  - Avellino
  - Milan
  - Roma
  - Torino
  - Viterbo
- Seoul, South Korea
- Spain (4):
  - Barcelona
  - Madrid
  - Málaga
  - Seville
- Taiwan (2):
  - Kaohsiung City
  - Taipei
- Nassau, The Bahamas
- Ukraine (4):
  - Dnipropetrovsk
  - Donetsk
  - Uzhhorod
  - Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aveo Pharmaceuticals, Inc. official web page — http://aveooncology.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the inclusion and none of the exclusion criteria were enrolled
Pre-assignment Details: All participants underwent inclusion and exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study related procedures.
  The study was terminated prior to completing enrollment, hence descriptive statistical analyses were performed for a limited set of data.
Groups:
- Placebo in Combination With Paclitaxel: Participants received placebo orally once daily with 90 mg/m2 of paclitaxel administered intravenously beginning on Day 1 for 3 weeks followed by 1 week off treatment.
- Tivozanib Hydrochloride in Combination With Paclitaxel: Participants received 1.5 mg tivozanib hydrochloride orally once daily with 90 mg/m2 of paclitaxel administered intravenously beginning on Day 1 for 3 weeks followed by 1 week off treatment.
Period: Overall Study
Arm/Group | Placebo in Combination With Paclitaxel | Tivozanib Hydrochloride in Combination With Paclitaxel
Started | 8 | 22
Treated | 8 | 21
Completed | 0 | 0
Not Completed | 8 | 22
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Termination of The Study by The Sponsor | 6 | 18
Not completed — Other Reasons Unspecified | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo in Combination With Paclitaxel | Tivozanib Hydrochloride in Combination With Paclitaxel | Total
Number analyzed (Participants) | 8 | 22 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 20 | 24
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (16.02) | 54.5 (10.06) | 56.3 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 22 | 30
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 14 | 22
  Black | 0 | 5 | 5
  Asian | 0 | 2 | 2
  Dominican | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (10.67) | 182.3 (708.53) | 144.4 (613.48)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Progression-free Survival (PFS) of Subjects
Description: PFS is defined as the time from randomization to progressive disease (PD) or death. The PFS comparison was performed for subjects treated with tivozanib hydrochloride in combination with paclitaxel vs placebo in combination with paclitaxel.
Time Frame: approximately 24 months
Population: The study was terminated prior to completing enrollment; due to low enrollment, no data was collected for this outcome measure.
Groups:
- Tivozanib Hydrochloride in Combination With Paclitaxel: 1.5 mg tivozanib hydrochloride orally once daily for 3 weeks followed by 1 week off and 90 mg/m2 of paclitaxel administered intravenously on weeks 1, 2 and 3 (Day 1, Day 8 and Day 15) of a 4-week cycle.
- Placebo in Combination With Paclitaxel: Placebo orally once daily for 3 weeks followed by 1 week off and 90 mg/m2 of paclitaxel administered intravenously on weeks 1, 2 and 3 (Day 1, Day 8 and Day 15) of a 4-week cycle.
Arm/Group | Tivozanib Hydrochloride in Combination With Paclitaxel | Placebo in Combination With Paclitaxel
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Comparison of Objective Response Rate (ORR) and Duration of Response (DoR) of Subjects
Description: ORR is defined as the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period. DoR is defined as the length of time that a tumor continues to respond to treatment without the cancer growing or spreading. The ORR and DoR comparison was performed for subjects treated with tivozanib hydrochloride in combination with paclitaxel vs placebo in combination with paclitaxel.
Time Frame: approximately 24 months
Population: as for outcome 1
Arm/Group | Tivozanib Hydrochloride in Combination With Paclitaxel | Placebo in Combination With Paclitaxel
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Comparison of Overall Survival (OS) of Subjects
Description: OS measures how long subjects, who undergo a certain treatment regimen, live compared to subjects who are in a control group (i.e., taking either another drug or an inactive treatment, known as a placebo). OS comparison was performed for subjects treated with tivozanib hydrochloride in combination with paclitaxel vs placebo in combination with paclitaxel.
Time Frame: approximately 24 months
Population: as for outcome 1
Arm/Group | Tivozanib Hydrochloride in Combination With Paclitaxel | Placebo in Combination With Paclitaxel
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Safety and Tolerability of Tivozanib Hydrochloride in Combination With Paclitaxel vs Placebo in Combination With Paclitaxel
Description: Number of subjects with serious and non-serious adverse events.
Time Frame: approximately 24 months
Population: Descriptive statistical analyses were performed for a limited set of data (disposition, demographics, and adverse events).
Measure: Count of Participants; unit: Participants
Arm/Group | Tivozanib Hydrochloride in Combination With Paclitaxel | Placebo in Combination With Paclitaxel
Number analyzed (Participants) | 21 | 8
Participants
  Subjects with serious adverse events | 1 | 1
  Subjects with non-serious adverse events | 19 | 8

5. Secondary Outcome: Pharmacokinetics (PK) of Tivozanib Hydrochloride and Paclitaxel When Administered in Combination
Description: PK is defined as the study of the bodily absorption, distribution, metabolism, and excretion of drugs.
Time Frame: approximately 24 months
Population: as for outcome 1
Arm/Group | Tivozanib Hydrochloride in Combination With Paclitaxel | Placebo in Combination With Paclitaxel
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Identification of Hypoxia Gene Signature
Description: Evaluation of hypoxia gene signature as a predictive biomarker of tivozanib hydrochloride response and establish the optimal cut-off to identify biomarker positive and negative subgroups. The genes comprising the hypoxia gene signature was analyzed in tumor tissue from subjects.
Time Frame: Cycle 1, Day 1: Pre-dose and 2, 4 and 24 hours post dose; Cycle 1, Day 8: Pre-dose; Cycle 1, Day 21: Pre-dose and 2, 4, 24, 48, and 96 hours post dose; Cycle 2 (Day 1): Pre-dose
Population: as for outcome 1
Arm/Group | Tivozanib Hydrochloride in Combination With Paclitaxel | Placebo in Combination With Paclitaxel
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Measurement of Subjects' Quality of Life (QoL)
Description: The Functional Assessment of Cancer Therapy-Breast (FACT-B) and Euro Quality of Life - 5 Dimensions (EQ-5D) questionnaires was used throughout the study to measure subjects' health-related QoL.
Time Frame: approximately 24 months
Population: as for outcome 1
Arm/Group | Tivozanib Hydrochloride in Combination With Paclitaxel | Placebo in Combination With Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 months
Description: Serious treatment-emergent adverse events and treatment emergent adverse events in Safety Population was reported.
Arm/Group | Placebo in Combination With Paclitaxel | Tivozanib Hydrochloride in Combination With Paclitaxel
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/21
Other Adverse Events (participants affected / at risk) | 8/8 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo in Combination With Paclitaxel (N=8) | Tivozanib Hydrochloride in Combination With Paclitaxel (N=21)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo in Combination With Paclitaxel (N=8) | Tivozanib Hydrochloride in Combination With Paclitaxel (N=21)
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 7
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis Genralized (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 9
Constipation (Gastrointestinal disorders) | 3 | 6
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 6
Vomiting (Gastrointestinal disorders) | 1 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 2
Faitgue (General disorders) | 4 | 11
Oedema peripheral (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 3
Platelet count increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 3
Lipase increased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 4
Dysgeusia (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 1 | 4
Neuropathy peripheral (Nervous system disorders) | 1 | 5
Presyncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Rash pustular (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Poor venous access (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 7
Endocrine disorders (Endocrine disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The Sponsor terminated Study AV-951-12-204 before enrollment was completed after determining that enrollment of subjects was much lower than expected, and that timely completion of the study was not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No